CLINICAL TRIAL: NCT01432548
Title: Ischemic Preconditioning Versus Intermittent Portal Triad Clamping in Liver Resection. Prospective Randomized Comparison
Brief Title: Ischemic Preconditioning. Prospective Comparison
Acronym: IP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Agudos "Dr. Cosme Argerich" (Other)
Responsible Party: Principal Investigator, Juan Marcelo Rivaldi, Ischemic preconditioning vs intermittent portal triad clamping in liver resection. Prospective Randomized Comparison, Hospital General de Agudos "Dr. Cosme Argerich"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JLendoire2
Record Dates: First submitted 2011-08-29; First posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Ischemic Lesions
Keywords: Ischemic; preconditioning; liver; resection
MeSH Terms: conditions — Ischemia | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: ischemic preconditioning — Surgery with ischemic preconditioning in liver resection

SUMMARY:
Vascular occlusion is used to reduce blood loss during liver resection (LR), but may cause ischemic damage to the remnant liver and can lead to liver failure in case of chronic liver disease. This restriction of blood flow (ischemia) and subsequent restoration (reperfusion) causes a harm that is called ischemia- reperfusion injury. Injuries sustained during the ischemic phase are related to a lack of oxygen to reduce cellular respiratory events can lead to, in a few minutes, irreversible damage. Ischemic preconditioning as a technique to protect the liver parenchyma during liver resection consists of an initial flow clamping for 10 minutes, with subsequent reperfusion for 10-15min, followed by a complete portal triad clamping during transection.

DETAILED DESCRIPTION:
Detailed Description:

This is a prospective controlled trial, conducted between July 2011 and July 2012. This study has been initiated by Liver & Transplant Division, Hospital Dr Cosme Argerich, Buenos Aires Argentina. The protocol was approved by ethics committees and an informed consent was obtained from each patient before they were enrolled. Sixty patients were randomized to either receive ischemic preconditioning prior to liver resection under intermittent pedicle clamping or Intermittent Pringle ischemia. Ischemic preconditioning was performed through a sequence of 10 minutes vascular inflow occlusion and 10 minutes of reperfusion prior to continuous pedicle clamping during resection. Intermittent pedicle clamping was conducted through a sequence of 15 minutes of vascular inflow occlusion and 5 minutes of reperfusion. The randomization process which was centralized was held in the operating room after inclusion criteria had been check and exclusion criteria ruled out.

ELIGIBILITY:
Inclusion Criteria:

* patients' age ≥ 18 years old
* Portal vein embolization allowed

Exclusion Criteria:

* laparoscopic liver resection
* pregnant women
* lack of patient consent
* lack of acceptance of the operating surgeon
* Hilar cholangiocarcinoma
* Simultaneous hepaticojejunostomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Mortality Complications | within 30 days after surgery

SECONDARY OUTCOMES:
Operative variables,markers of liver function and injury, pathological parenchymal characteristics | within 30 days after surgey
  Operative time Transection time Operative blood loss Transection area Intraoperative haemodynamic and gases parameters (CVP, MAP) Requirement of blood products. ICU and total length of hospital stay Markers of liver function (Bilirrubin, prothtrombin time) Markers of liver injury (aspartate aminotransferase (AST), alanine aminotransferase (ALT) Pathological parenchymal characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Dr Cosme Argerich, Buenos Aires, Buenos Aires, Argentina